CLINICAL TRIAL: NCT05051748
Title: Clinical Evaluation of Different Minimal Invasive Treatment Modalities of Mild to Moderate Dental Fluorosis Using A Visual Analog Scale
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Mostafa Nasser Abdelmoniem Youssef, Mostafa Nasser Abdelmoniem Youssef, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202/2019
Record Dates: First submitted 2021-09-11; First posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Dental Fluorosis
Keywords: Bleaching, microabrasion, CPP-ACFP, VAS
MeSH Terms: conditions — Fluorosis, Dental | interventions — opalustre

STUDY DESIGN:
Intervention Model Description: Fluorosed teeth
Who Masked: Participant, Investigator
Masking Description: Masking was ensured as the baseline and follow-ups photographs were stored on a computer with a unique ID and the investigators were not disclosed about the participants' treatment protocol. Blinding of the participants was guaranteed as they didn't know each other, or the treatments received in other protocols
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- In-office bleaching (Active Comparator): 40% hydrogen peroxide in-office bleaching (Opalescence™ boost™ PF 40%, Ultradent Products, Inc., South Jordan, UT, USA)
  Interventions: Other: Opalescence™ boost™ PF 40%
- microabrasion (Active Comparator): 6.6% hydrochloric acid and silicon carbide microparticles microabrasion paste (Opalustre™, Ultradent Products, Inc., South Jordan, UT, USA).
  Interventions: Other: Opalustre™
- Remineralization (Active Comparator): casein phosphopeptide amorphous calcium fluoride phosphate (CPP-ACFP) remineralizing tooth crème (MI-Paste Plus®, GC America Inc., USA).
  Interventions: Other: MI-Paste Plus®
- Microabrasion + In-office bleaching (Active Comparator): teeth were treated with enamel microabrasion followed by in-office bleaching.
  Interventions: Other: Opalescence™ boost™ PF 40%; Other: Opalustre™
- In-office bleaching + Remineralization (Active Comparator): n-office bleaching was applied followed by MI-Paste Plus®
  Interventions: Other: Opalescence™ boost™ PF 40%; Other: MI-Paste Plus®
- Microabrasion + Remineralization (Active Comparator): microabrasion was applied followed by MI-Paste Plus®
  Interventions: Other: Opalustre™; Other: MI-Paste Plus®
- Microabrasion + In-office bleaching + Remineralization (Active Comparator): teeth were treated with microabrasion followed by in-office bleaching and lastly MI-Paste Plus®
  Interventions: Other: Opalescence™ boost™ PF 40%; Other: Opalustre™; Other: MI-Paste Plus®
- Control (No Intervention): no treatment (control).

INTERVENTIONS:
Other: Opalescence™ boost™ PF 40% — 40% hydrogen peroxide in-office bleaching
  Arms: In-office bleaching; In-office bleaching + Remineralization; Microabrasion + In-office bleaching; Microabrasion + In-office bleaching + Remineralization
Other: Opalustre™ — 6.6% hydrochloric acid and silicon carbide microparticles microabrasion paste
  Arms: Microabrasion + In-office bleaching; Microabrasion + In-office bleaching + Remineralization; Microabrasion + Remineralization; microabrasion
Other: MI-Paste Plus® — casein phosphopeptide amorphous calcium fluoride phosphate (CPP-ACFP) remineralizing tooth crème
  Arms: In-office bleaching + Remineralization; Microabrasion + In-office bleaching + Remineralization; Microabrasion + Remineralization; Remineralization

SUMMARY:
This study was conducted for clinical evaluation of the quality of different minimal-invasive treatment modalities and combination treatments in esthetics improvement of mild to moderate fluorosed teeth using two different evaluation methods.

One hundred and sixty fluorosed teeth were included in this study. Prior to the interventions, pre-operative photographs were taken as baseline records. After that teeth were randomly allocated in eight treatment protocols with twenty teeth (n=20) included in each protocol. Protocol one (P1) Opalescence™ boost™ PF 40%. Protocol two (P2) Opalustre™. Protocol three (P3) MI-Paste Plus®. In protocol four (P4) teeth were treated with Opalustre™ followed by Opalescence™ boost™ PF 40%. In protocol five (P5) Opalescence™ boost™ PF 40% was applied followed by MI-Paste Plus®, while in protocol six (P6) Opalustre™ was applied followed by MI-Paste Plus®. Whereas protocol seven (P7) teeth were treated with Opalustre™ followed by Opalescence™ boost™ PF 40% and lastly MI-Paste Plus®. Protocol eight (P8) control.

All teeth were evaluated immediately after treatment (T1), after 14 days (T2), after 3 months (T3) and after 6 months (T4).

They were rated for "improvement in appearance" and "change in white/brown opaque areas" using VAS through two blinded evaluators by comparing photographs of each follow-up time point with baseline. "Patient satisfaction", "tooth sensitivity" and "requirements for further treatments" were recorded by the participant.

DETAILED DESCRIPTION:
This study was conducted for clinical evaluation of the quality of different minimal-invasive treatment modalities and combination treatments in esthetics improvement of mild to moderate fluorosed teeth using two different evaluation methods.

Materials used in this study were Opalustre™ (microabrasion paste of 6.6% hydrochloric acid and Silicon Carbide), Opalescence™ Boost™ PF 40% (in-office bleaching of 40% hydrogen peroxide) and MI-Paste Plus® (topical remineralizing tooth crème of casein phosphopeptide amorphous calcium fluoride phosphate).

One hundred and sixty fluorosed teeth were included in this study. Prior to the interventions, pre-operative photographs were taken as baseline records. After that teeth were randomly allocated in eight treatment protocols with twenty teeth (n=20) included in each protocol. Protocol one (P1) Opalescence™ boost™ PF 40%. Protocol two (P2) Opalustre™. Protocol three (P3) MI-Paste Plus®. In protocol four (P4) teeth were treated with Opalustre™ followed by Opalescence™ boost™ PF 40%. In protocol five (P5) Opalescence™ boost™ PF 40% was applied followed by MI-Paste Plus®, while in protocol six (P6) Opalustre™ was applied followed by MI-Paste Plus®. Whereas protocol seven (P7) teeth were treated with Opalustre™ followed by Opalescence™ boost™ PF 40% and lastly MI-Paste Plus®. Protocol eight (P8) control.

All teeth were evaluated immediately after treatment (T1), after 14 days (T2), after 3 months (T3) and after 6 months (T4).

They were rated for "improvement in appearance" and "change in white/brown opaque areas" using VAS through two blinded evaluators by comparing photographs of each follow-up time point with baseline. "Patient satisfaction", "tooth sensitivity" and "requirements for further treatments" were recorded by the participant.

Data were collected, checked, revised and organized in tables and figures using Microsoft Excel 2016.Improvement in appearance, change in opacity, tooth sensitivity, patient satisfaction and requirement for further treatment were not normally distributed (p<0.05*) i.e. nonparametric data, accordingly, Freidman's test to differentiate between timepoints and Kruskal-Wallis to compare between treatment protocols were applied at 0.05 level.

ELIGIBILITY:
Inclusion Criteria:

* Each participant had at least 8 teeth with mild to moderate dental fluorosis score 1-4 according to Thylstrup and Fejerskov index.
* Participants of age range 20-35 years old
* Good oral and general health
* Had no caries or restorations on the teeth to be treated
* Ability to return for periodic recalls

Exclusion Criteria:

* Hypersensitive teeth
* Any fixed orthodontic appliance
* Current or previous use of bleaching agents
* A history of allergies to tooth whitening product
* Smoking habits
* Pregnant or lactating women
* Non-vital or teeth with symptoms of pulpitis
* Loss or fracture of maxillary and mandibular anterior teeth

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-08 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | Six Months
  Participants were asked to score for "patient satisfaction" using VAS ranging from 1 to 7

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Suez canal university, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No